CLINICAL TRIAL: NCT02211612
Title: Role of Fatty Acids in Skeletal Muscle Hypertrophy and Ectopic Fat Accumulation During Overfeeding (LIPOGAIN-2)
Brief Title: Overeating Different Fats and Influence on Muscle Mass and Body Fat Accumulation
Acronym: LIPOGAIN-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, David Iggman, MD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LIPOGAIN-2
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Overfeeding; Muscle Mass; Body Composition; Ectopic Fat
Keywords: Overfeeding; Weight gain; Liver fat; Pancreatic fat; Ectopic fat; Skeletal muscle; Adipose tissue; Gene expression; DNA methylation; Palmitate; Linoleic acid; Saturated fat; Polyunsaturated fat; Metabolism; Insulin sensitivity
MeSH Terms: conditions — Obesity; Weight Gain; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saturated fatty acids (SFA)-group (Experimental): Weight gain created by addition of muffins baked on saturated fat
  Interventions: Dietary Supplement: SFA-group
- Polyunsaturated fatty acids (PUFA)-group (Experimental): Weight gain created by addition of muffins baked on polyunsaturated fat
  Interventions: Dietary Supplement: PUFA-group

INTERVENTIONS:
Dietary Supplement: PUFA-group
  Arms: Polyunsaturated fatty acids (PUFA)-group
Dietary Supplement: SFA-group
  Arms: Saturated fatty acids (SFA)-group

SUMMARY:
To investigate metabolic and molecular response to fatty acid-specific overfeeding in overweight subjects, in relation to changes in ectopic fat, lean tissue mass and insulin sensitivity

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25-32

Exclusion Criteria:

* Type 2 diabetes
* Type 1 diabetes
* Kidney disease
* Liver disease
* Abnormal clinical chemistry at screening
* Intense physical exercise > 2 hours per week
* Use of statins or drugs affecting energy metabolism
* Use of extreme diets

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in lean tissue mass | 10 weeks
  Assessed by magnetic resonance imaging (MRI) and air displacement plethysmography (BodPod)

SECONDARY OUTCOMES:
Change in hepatic fat content | 10 weeks
  Assessed by magnetic resonance imaging (MRI)
Change in visceral adipose tissue (VAT) | 10 weeks
  Assessed by magnetic resonance imaging (MRI)
Change in total adipose tissue | 10 weeks
  Assessed by magnetic resonance imaging (MRI)
Change in pancreatic fat | 10 weeks
  Assessed by MRI
Change in insulin sensitivity | 10 weeks
  Assessed by oral glucose tolerance test (OGTT)
Change in plasma lipids | 10 weeks
  Plasma cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides, apolipoprotein B, apolipoprotein A1, free fatty acids, glycerol, proprotein convertase subtilisin/kexin type 9
Change in circulating inflammation and coagulation markers | 10 weeks
  Plasma tumor necrosis factor-receptor 2, Interleukin receptor 1 antagonist, C-reactive protein, fibrinogen, adhesion molecules

OTHER OUTCOMES:
Circulating hormones and molecular analyses in muscle and fat tissue | 10 weeks
  Serum hormones including prolactin, tyroxin, T3, cortisol, growth hormone, Insulin growth factor-1. Fat cell morphology assessment in fat tissue, and gene and protein expression, DNA methylation analyses in fat and muscle tissue, palmitate tracer uptake in liver using positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Riserus, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University; Clinical nutrition and metabolism; Dept of public health and caring sciences, Uppsala, Please Select, Sweden

REFERENCES:
- [Derived] Rosqvist F, Cedernaes J, Martinez Mora A, Friden M, Johansson HE, Iggman D, Larsson A, Ahlstrom H, Kullberg J, Riserus U. Overfeeding polyunsaturated fat compared with saturated fat does not differentially influence lean tissue accumulation in individuals with overweight: a randomized controlled trial. Am J Clin Nutr. 2024 Jul;120(1):121-128. doi: 10.1016/j.ajcnut.2024.04.010. Epub 2024 Apr 16. PMID 38636844
- [Derived] Rosqvist F, Orho-Melander M, Kullberg J, Iggman D, Johansson HE, Cedernaes J, Ahlstrom H, Riserus U. Abdominal Fat and Metabolic Health Markers but Not PNPLA3 Genotype Predicts Liver Fat Accumulation in Response to Excess Intake of Energy and Saturated Fat in Healthy Individuals. Front Nutr. 2020 Dec 3;7:606004. doi: 10.3389/fnut.2020.606004. eCollection 2020. PMID 33344496
- [Derived] Rosqvist F, Kullberg J, Stahlman M, Cedernaes J, Heurling K, Johansson HE, Iggman D, Wilking H, Larsson A, Eriksson O, Johansson L, Straniero S, Rudling M, Antoni G, Lubberink M, Orho-Melander M, Boren J, Ahlstrom H, Riserus U. Overeating Saturated Fat Promotes Fatty Liver and Ceramides Compared With Polyunsaturated Fat: A Randomized Trial. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6207-6219. doi: 10.1210/jc.2019-00160. PMID 31369090